CLINICAL TRIAL: NCT06297070
Title: Promoting ReprOductive WellbEing Through Shared Medical Appointments and Health Coaching Sessions
Brief Title: Lifestyle Care for Fertility Outcome Evaluation
Acronym: PROWESS
Status: Completed | Type: Observational
Sponsor: Christine Kaiser, LAc, DACM (Other)
Responsible Party: Sponsor-Investigator, Christine Kaiser, LAc, DACM, Principal Investigator, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Other Study IDs: STUDY20231406
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Fertility Issues
Keywords: fertility; shared medical appointments; health coaching; quality of life
MeSH Terms: conditions — Infertility | interventions — Fertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Whole Health Lifestyle Care for Reproductive Well-being pilot program — The program consists of an individual Integrative Health and Medicine (IHM) consultation with a CWH IHM provider, 4 Shared Medical Appointments (SMA), and 4 individual Health and Wellness Coaching (HWC) sessions. The SMA sessions occur at the UH CWH Beachwood office conference and movement rooms. The HWC sessions are virtual. The consultations are either virtual or in person at UH CWH Beachwood.
  Other Names: Lifestyle Care for Fertility

SUMMARY:
An observational outcome evaluation of the Lifestyle Care for Fertility program.

DETAILED DESCRIPTION:
This outcome evaluation will examine the feasibility and acceptability of the Whole Health Lifestyle Care for Reproductive Well-being Pilot Program ("Lifestyle Care for Fertility" or LCF) and collection of health behavior and patient-reported outcomes. Secondarily, it will also examine the longitudinal changes in health behaviors and patient-reported outcomes of participants in the Lifestyle Care for Fertility program

The Lifestyle Care for Fertility program serves women who have a fertility-related diagnosis. The program consists of an individual Integrative Health and Medicine (IHM) consultation with a CWH IHM provider, 4 Shared Medical Appointments (SMA), and 4 individual Health and Wellness Coaching (HWC) sessions. The SMA sessions occur at the UH CWH Beachwood office conference and movement rooms. The HWC sessions are virtual. The consultations are either virtual or in person at UH CWH Beachwood. Topics include meditation, sleep, yoga/exercise/movement, acupuncture, and nutrition

Participation in the program is not contingent on participation in the outcome evaluation. Patients with a uterus aged 18-50 who have a fertility-related diagnosis are eligible to participate in the program. Participants in the outcome evaluation will be a subset of the participants in the program who give their consent to researchers to collect survey and EHR data.

The outcome evaluation will collect data at 4 weeks, 8 weeks, and before, after, and in between each of the 8 weekly sessions. Data collected at baseline include demographics, PROMIS Sleep Disturbance 8a, Perceived Stress Scale 4 (PSS-4), Infertility Self Efficacy Scale (ISE), and current Health Behaviors (HB). The HB survey will be administered between Sessions 1-8, as well as after Session 8, to observe any longitudinal changes. Patients will complete the PROMIS Sleep Disturbance 8a, PSS-4, and ISE at 4 weeks and 8 weeks. Pre- and post-session data includes 0-10 NRS ratings of stress, energy, focus, well-being, perceived support (post-only), and satisfaction (post-only). Additionally, participants will complete a satisfaction survey post Session 8. All data will be collected in REDCap via a text message or email link sent to the participant. Research staff will review the participant's medical record to collect data on the participant's demographics and clinical characteristics at baseline, and to collect chemical pregnancy data at six months after the 8 sessions have been completed. Attendance data about participants will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult with a uterus aged from 18 to 50 years
* Participating in the Lifestyle Care for Fertility program
* Able to speak and understand English.
* Has email address and access to mobile device with a functioning data plan.
* Infertility-related diagnosis

Exclusion Criteria:

* Age < 18 or > 50 years
* Having a significant and uncorrected visual, hearing, or cognitive impairment
* Inability to provide consent
* Current pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study participants will be patients of University Hospitals Connor Whole Health who have a fertility-related diagnosis and who are participating in the Lifestyle Care for Fertility program
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Servings of Fruit | 8 weeks
  Number of servings of fruit consumed each day. A serving is about 1 medium piece, or 1/2 cup of fruit.
Servings of Vegetables | 8 weeks
  Number of servings of vegetables consumed each day. A serving is about 1 cup of raw leafy vegetables, 1/2 cup of other cooked or raw vegetables, or 3/4 cup of raw vegetable juice.
Glasses of Water | 8 weeks
  Number of glasses (8 oz) of plain water consumed per day.
Caffeinated Beverages | 8 weeks
  Number of caffeinated beverages consumed per day.
Aerobic Exercise | 8 Weeks
  Frequency of aerobic exercise (min 20 min) in last week.
Strengthening Exercise | 8 weeks
  Frequency of muscle strengthening exercise (min 20 min) in last week.
Stretching Exercise | 8 weeks
  Frequency of stretching exercise in last week.
Sleep Hygiene | 8 weeks
  Frequency of sleep hygiene practices before bed in last week.
Hours of Sleep | 8 weeks
  Average number of hours of sleep per night in last week.
Self Care - Biofeedback | 8 weeks
  Frequency of use of biofeedback in last week.
Self Care - Breathing Exercises | 8 weeks
  Frequency of breathing exercise practice in last week.
Self Care - Guided Imagery | 8 weeks
  Frequency of guided imagery practice in last week.
Self Care - Mindfulness/Meditation | 8 weeks
  Frequency of mindfulness/meditation practice in last week.
Self Care - Progressive Relaxation | 8 weeks
  Frequency of progressive relaxation practice in last week.
Self Care - Journaling/Gratitude Journaling | 8 weeks
  Frequency of journaling or gratitude journaling in last week.
Self Care - Tai Chi/Chi Gong | 8 weeks
  Frequency of Tai Chi or Chi Gong practice in last week.
Self-Care - Massage Therapy | 8 weeks
  Frequency of receipt of massage therapy in last week.
Self Care - Acupuncture/Acupressure | 8 weeks
  Frequency of receipt of acupuncture or acupressure in last week.
Self Care - Nature Walking | 8 weeks
  Frequency of walking in nature in last week.

SECONDARY OUTCOMES:
PROMIS Sleep Disturbance 8a | 8 weeks
  Composite score (8 -40 with higher scores representing a better outcome) measuring self-reported alertness, sleepiness, tiredness, and functional impairments associated with sleep problems during waking hours within the past seven days.
Perceived Stress Scale - 4 | 8 weeks
  Composite score (0-16 with higher scores representing a better outcome) measuring self-reported perception of stress.
Infertility Self Efficacy | 8 weeks
  Composite score (16-144 with higher scores representing a better outcome) measuring self-reported perceived self-efficacy for coping with a diagnosis and treatment for infertility.
Chemical pregnancy | 8 months
  Pregnancy as confirmed by presence of human chorionic gonadotropin (hCG) within 6 months of program completion.
Stress Change (level of stress: none [0] to worst possible [10]) - SMA | 2 hours
  Change in 11 point numerical rating scale. Range from -11 to 11, with lower scores representing better outcomes: Change in stress level from pre to post each of the 4 shared medical appointment sessions.
Anxiety Change (level of anxiety right now: none [0] to worst possible [10]) - SMA | 2 hours
  Change in 11 point numerical rating scale. Range from -11 to 11, with lower scores representing better outcomes: Change in anxiety level from pre to post each of the 4 shared medical appointment sessions.
Energy Change (level of energy right now: no energy [0] to most energized [10]) - SMA | 2 hours
  Change in 11 point numerical rating scale. Range from -11 to 11, with higher scores representing better outcomes: Change in energy level from pre to post each of the 4 shared medical appointment sessions.
Focus Change (level of energy right now: not focused at all [0] to very focused [10]) - SMA | 2 hours
  Change in 11 point numerical rating scale. Range from -11 to 11, with higher scores representing better outcomes: Change in focus level from pre to post each of the 4 shared medical appointment sessions.
Wellbeing Change (level of energy right now: worst possible [0] to best possible [10]) - SMA | 2 hours
  Change in 11 point numerical rating scale. Range from -11 to 11, with higher scores representing better outcomes: Change in wellbeing level from pre to post each of the 4 shared medical appointment sessions.
Stress Change (level of stress: none [0] to worst possible [10]) - HWC | 45 minutes
  Change in 11 point numerical rating scale. Range from -11 to 11, with lower scores representing better outcomes:
  Change in stress level from pre to post each of the 4 health and wellness coaching sessions.
Anxiety Change (level of anxiety right now: none [0] to worst possible [10]) - HWC | 45 minutes
  Change in 11 point numerical rating scale. Range from -11 to 11, with lower scores representing better outcomes: Change in anxiety level from pre to post each of the 4 health and wellness coaching sessions.
Energy Change (level of energy right now: no energy [0] to most energized [10]) - HWC | 45 minutes
  Change in 11 point numerical rating scale. Range from -11 to 11, with higher scores representing better outcomes: Change in energy level from pre to post each of the 4 health and wellness coaching sessions.
Focus Change (level of energy right now: not focused at all [0] to very focused [10]) - HWC | 45 minutes
  Change in 11 point numerical rating scale. Range from -11 to 11, with higher scores representing better outcomes: Change in focus level from pre to post each of the 4 health and wellness coaching sessions.
Wellbeing Change (level of energy right now: worst possible [0] to best possible [10]) - HWC | 45 minutes
  Change in 11 point numerical rating scale. Range from -11 to 11, with higher scores representing better outcomes: Change in wellbeing level from pre to post each of the 4 health and wellness coaching sessions.
Recruitment Rate | 4-6 weeks
  Number enrolled over number approached.
Retention Rate | 8 weeks
  Percent of participants retained at each data collection point
Pace of Accrual | 8 weeks
  Number of participants enrolled from each program cohort.
Data Completeness | 8 weeks
  Percent of data collection that is completed
Helpfulness of group sessions in addressing needs | 8 weeks
  5-point Likert scale strongly disagree to strongly agree (1 - 5 with higher scores representing better outcomes)
Coverage of important issues in the sessions | 8 weeks
  5-point Likert scale strongly disagree to strongly agree (1 - 5 with higher scores representing better outcomes)
Helpfulness of tools presented in nutrition session | 8 weeks
  5-point Likert scale strongly disagree to strongly agree (1 - 5 with higher scores representing better outcomes)
Helpfulness of tools presented in movement session | 8 weeks
  5-point Likert scale strongly disagree to strongly agree (1 - 5 with higher scores representing better outcomes)
Helpfulness of tools presented in relaxation and sleep session | 8 weeks
  5-point Likert scale strongly disagree to strongly agree (1 - 5 with higher scores representing better outcomes)
Helpfulness of tools presented in integrate session | 8 weeks
  5-point Likert scale strongly disagree to strongly agree (1 - 5 with higher scores representing better outcomes)
Enjoyed group sessions | 8 weeks
  5-point Likert scale strongly disagree to strongly agree (1 - 5 with higher scores representing better outcomes)
Enjoyed health and wellness coaching session | 8 weeks
  5-point Likert scale strongly disagree to strongly agree (1 - 5 with higher scores representing better outcomes)
Group setting was beneficial | 8 weeks
  5-point Likert scale strongly disagree to strongly agree (1 - 5 with higher scores representing better outcomes)
Comfortable in group setting | 8 weeks
  5-point Likert scale strongly disagree to strongly agree (1 - 5 with higher scores representing better outcomes)
Helpfulness of individual health coaching sessions | 8 weeks
  5-point Likert scale strongly disagree to strongly agree (1 - 5 with higher scores representing better outcomes)
Feedback questionnaire: Location Preference question 1 | 8 weeks
  Shared Medical Appointment session location preference. Choices: virtual, in person or no preference.
Feedback questionnaire: Location Preference question 2 | 8 weeks
  Health and Wellness Coaching session location preference. Choices: virtual, in person or no preference.
Feedback questionnaire: Number of Sessions question. | 8 weeks
  Opinion on number of sessions. Choices: too few, just right, too many.
Feedback questionnaire: Length of Sessions question. | 8 weeks
  Opinion on length of sessions. Choices: too short, just right, too long.
Rating of level of support during each SMA | 2 hours
  11-point Likert scale not supported to very well supported (0 - 10 with higher scores representing better outcomes): Level of support received during each of the 4 shared medical appointment sessions.
Rating of level of support during HWC | 45 minutes
  11-point Likert scale not supported to very well supported (0 - 10 with higher scores representing better outcomes): Level of support received during each of the 4 health and wellness coaching sessions.
Overall level of satisfaction during each SMA | 2 hours
  11-point Likert scale not at all satisfied to very well satisfied (0 - 10 with higher scores representing better outcomes): Overall level of satisfaction with each of the 4 shared medical appointment sessions.
Overall level of satisfaction during each HWC | 45 minutes
  11-point Likert scale not at all satisfied to very well satisfied (0 - 10 with higher scores representing better outcomes): Overall level of satisfaction with each of the 4 health and wellness coaching sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Kaiser, DACM LAc, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT06297070/Prot_SAP_000.pdf